CLINICAL TRIAL: NCT01683994
Title: A Phase I and Randomized Phase II Multicenter Study of Cabozantinib (XL184) Plus Docetaxel and Prednisone in Metastatic Castrate Resistant Prostate Cancer
Brief Title: Cabozantinib Plus Docetaxel and Prednisone for Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Dahut Jr., M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120204; 12-C-0204
Record Dates: First submitted 2012-09-08; First posted 2012-09-12 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Prostatic Neoplasms
Keywords: Angiogenesis Inhibitors; Small Molecules; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- combination of cabozantinib, docetaxel and prednisone (Experimental): combination of cabozantinib, docetaxel and prednisone
  Interventions: Drug: Cabozantinib; Drug: Docetaxel; Drug: Prednisone
- PII/ Arm 1-docetaxel + prednisone only (Active Comparator): docetaxel + prednisone only
  Interventions: Drug: Docetaxel; Drug: Prednisone
- PII/Arm 2 -docetaxel+ prednisone + cabozantinib (Active Comparator): docetaxel+ prednisone + cabozantinib
  Interventions: Drug: Cabozantinib; Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Cabozantinib — Assigned dose given daily during each 21 day cycle. Treatment may continue until disease progression or intolerable toxicity.
  Other Names: Cometriq
  Arms: PII/Arm 2 -docetaxel+ prednisone + cabozantinib; combination of cabozantinib, docetaxel and prednisone
Drug: Docetaxel — 75mg/m^2 intravenous (IV) over approximately 60 minutes on cycle 1 day 1 and repeated every 21 days until disease progression or intolerable toxicity.
  Other Names: Taxotere
Drug: Prednisone — 5 mg by mouth (PO) twice a day during each 21 day cycle until disease progression or intolerable toxicity.
  Other Names: Deltasone

SUMMARY:
Background:

- Cabozantinib is a drug that slows the growth of blood vessels that feed tumors. It is approved for medullary thyroid cancer. However, studies have shown that prostate tumors respond to it. Docetaxel and prednisone are standard treatments for advanced prostate cancer. Researchers want to see if adding cabozantinib to these two drugs can be a safe and effective treatment for this type of cancer.

Objectives:

- To test the safety and effectiveness of cabozantinib with standard treatments for advanced prostate cancer.

Eligibility:

- Individuals at least 18 years of age who have advanced prostate cancer that has not responded to standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies will also be performed.
* Participants will receive the cancer drugs over 21-day cycles of treatment. They will take docetaxel and cabozantinib on day 1 of each cycle. Each docetaxel infusion will take about 1 hour. They will also take prednisone by mouth twice each day.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will continue to take the study drugs for as long as their cancer does not worsen and side effects are not too severe.

DETAILED DESCRIPTION:
Background:

* Docetaxel is established as first-line chemotherapy in patients with metastatic castrate resistant prostate cancer (CRPC). However; it is increasingly recognized that combining docetaxel with other agents of clinical activities without overlapping toxicities could simultaneously target different cellular signaling pathways vital for tumor survival, producing either additive or synergistic activities.
* Inhibition of angiogenesis, either as a stand-alone approach or in combination with chemotherapy, has demonstrable antitumor efficacy against CRPC and there are several antiangiogenic agents that are now in clinical trials in this population of patients.
* Cabozantinib (XL184) was developed as an inhibitor of both angiogenesis and of its resistance mechanism. It is an inhibitor of multiple receptor tyrosine kinases including tyrosine-protein kinase Met (c-Met), vascular endothelial growth factor receptor 2 (VEGFR2) and rearranged during transfection (RET).
* In single agent clinical studies, cabozantinib demonstrated, broad anti-tumor activities across many solid tumor types.

Objectives:

* To determine the safety profile of cabozantinib in combination with docetaxel and prednisone, and to determine the maximal tolerated dose (MTD) as recommended phase II dose in combination with docetaxel
* To determine the relative efficacy (in terms of progression free survival (PFS)) of docetaxel and cabozantinib compared to docetaxel alone

Eligibility:

* Patients must have progressive metastatic CRPC. There must be radiographic evidence of disease after primary treatment with surgery or radiotherapy. If patients had been on flutamide, they must have disease progression at least 4 weeks after withdrawal. Patients on bicalutamide or nilutamide must have progression at least 6 weeks after withdrawal. Withdrawal criteria apply only to patients on the above anti-androgens for at least the prior 6 months.
* Patients must be at least 18 years of age and able to give informed consent.
* Patients in the Phase II portion of the study must have progressed on abiraterone or enzalutamide

Design:

* The initial phase I portion of this study will test fixed dose docetaxel and prednisone in combination with cabozantinib at three escalating doses. Using a standard 3 + 3 design, three patients will initially be treated at each dose level until MTD has been defined.
* An expansion cohort will then be enrolled at the MTD to further characterize safety, toxicity and pharmacokinetic data and to obtain preliminary information on the efficacy of the combination treatment.
* In Phase II, patients will be enrolled to a randomized two-arm cohort comparing docetaxel in combination with cabozantinib to docetaxel alone with a primary endpoint of PFS.
* The accrual ceiling for the study, including the Phase I dose escalation and the expansion phases as well as the Phase II randomized phase, is set at 81.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Must have metastatic, progressive, castrate resistant prostate cancer (CRPC). There must be radiographic evidence of disease after primary treatment with surgery or radiotherapy that has continued to progress radiographically or biochemically (rising PSA levels on successive measurements) despite adequate androgen-deprivation therapy, which is defined as having undergone bilateral surgical castration or continued treatment on GnRH agonists or antagonists.

Progression must be evidenced and documented by any of the following parameters:

* Two consecutively rising PSA values, above the baseline, at a minimum of 1- week intervals
* Appearance of one or more new lesions on bone scan
* Progressive measurable disease by RECIST 1.1

The use of androgen receptor inhibitors is not required prior to study entry. For those patients receiving an anti-androgen agent (flutamide, bicalutamide, or nilutamide), for at least 6 consecutive months immediately prior to study entry, and are entering the trial due to a rise in PSA, they must demonstrate a continued rise in PSA within 4 weeks after stopping flutamide and within 6 weeks after stopping bicalutamide or nilutamide. Flutamide, nilutamide and bicalutamide disease progression requirements only apply to patients who have been on these drugs for at least the prior 6 months.

* Histopathological confirmation of prostate cancer by the Laboratory of Pathology of the National Cancer Institute (NCI) Pathology Department of the Walter Reed National Military Medical Center or YALE is required prior to entering this study. Patients whose pathology specimens are no longer available may be enrolled if the patient has a clinical course that is consistent with prostate cancer and available documentation from an outside pathology laboratory of the diagnosis. All efforts should be made to have the material forwarded to the research team for use in correlative studies in cases where original tissue blocks or archival biopsy material is available.
* Patients must have metastatic disease, defined as at least one lesion on bone scan or at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam.
* Patients must have a performance status of 0 to 2 according to the ECOG criteria.
* Patients must have adequate bone marrow, hepatic, and renal function with:

  * Hemoglobin greater than or equal to 9 grams per deciliter
  * Leukocytes greater than or equal to 3000 per microliters
  * ANC greater than or equal to 1500 per microliters, without CSF support
  * Platelets greater than or equal to 100,000 per microliters
  * AST (SGOT) less than or equal to 2.5 times upper limit of normal (ULN)
  * ALT (SGPT) less than or equal to 2.5 times upper limit of normal (ULN)
  * Total serum bilirubin less than or equal to the upper limit of normal (ULN)
  * Serum albumin greater than or equal to 2.8 grams per deciliters
  * Serum phosphorus, calcium, magnesium, and potassium greater than or equal to LLN
  * Lipase less than 2.0 times the upper limit of normal and no radiologic or clinical evidence of pancreatitis
  * Creatinine less than or equal to 1.5 times institutional upper limits of normal

OR

* creatinine clearance of greater than or equal to 50 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal by 24 hour urine.
* urine protein/urine creatinine ratio (UPCR) less than or equal to 1

  * Patients must be at least 18 years of age. Because no dosing or adverse event data are currently available on the use of cabozantinib in combination with docetaxel and prednisone in patients less than 18 years of age, children are excluded from this study, but may be eligible for future pediatric trials
  * Patient must be capable of understanding and complying with protocol requirements and is willing to give informed consent
  * Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of XL184 administration. Sexually active subjects and their female partners must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must also agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s). Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
  * Patients enrolled on the randomized portion of the study must have had disease progression on arbiraterone or enzalutamide.

EXCLUSION CRITERIA:

* The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment
* The subject is unable to swallow tablets
* The subject has tumor invading (or there is concern for invasion of) major blood vessel
* The subject has active brain metastases or epidural disease Subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible. Neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment. Baseline brain scans are not required to confirm eligibility.
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel). Low dose aspirin (less than or equal to 81 milligrams per day), low-dose warfarin (less than or equal to1 milligrams per day), and prophylactic low molecular weight heparin (LMWH) are permitted.
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) greater than 500 milliseconds within 28 days before initiation of protocol therapy. Note: if initial QTcF is found to be greater than 500 milliseconds, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is less than or equal to 500 milliseconds, the subject meets eligibility in this regard.
* Patients with contraindication to steroid use
* Prior treatment with cabozantinib
* The patient has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 3 weeks, or nitrosoureas or mitomycin within 6 weeks before the first dose of study treatment.
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment with the exception of patients receiving prior abiraterone or ketoconazole. For patients receiving prior abiraterone or ketoconazole, they must discontinue the medication within 5 half lives of the compound before the first dose of study treatment in order to participate in this study. Note: Subjects with prostate cancer currently receiving LHRH or GnRH agonists must be maintained on these agents.
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
* The subject has received radiation therapy:

  * to the thoracic cavity or gastrointestinal tract within 3 months before the first dose of study treatment
  * to bone or brain metastasis within 14 days before the first dose of study treatment
  * to any other site(s) within 28 days before the first dose of study treatment
* The subject has received radionuclide treatment within 6 weeks prior to the first dose of the study treatment
* The subject has not recovered to baseline or CTCAE less than or equal to Grade 1 from toxicity due to all prior therapies, including surgery, except alopecia and other non-clinically significant AEs.
* The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test results at screening greater than or equal 1.3 times the laboratory ULN within 7 days before the first dose of study treatment
* The subject has experienced any of the following:

  * clinically-significant hematemesis or gastrointestinal bleeding within 6 months before the first dose of study treatment
  * hemoptysis of greater than or equal to 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including

    * Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained BP greater than 140 millimeters of mercury systolic, or greater than 90 millimeters of mercury diastolic despite optimal antihypertensive treatment (BP must be controlled at screening)
    * Any history of congenital long QT syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * unstable angina pectoris
      * clinically-significant cardiac arrhythmias
      * stroke (including TIA, or other ischemic event)
      * myocardial infarction

        * thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following within 28 days before the first dose of study treatment

      * intra-abdominal tumor/metastases invading GI mucosa
      * active peptic ulcer disease
      * inflammatory bowel disease (including ulcerative colitis and Crohns disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis

        * malabsorption syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * history of abdominal fistula
      * gastrointestinal perforation
      * bowel obstruction or gastric outlet obstruction
      * intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months ago.
  * Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy or concurrent evidence of intraluminal tumor involving the trachea and esophagus.

    * Other clinically significant disorders such as:

      * active infection requiring intravenous treatment within 10 days of starting protocol
      * serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
      * history of organ transplant
      * concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
      * history of major surgery as follows:

        * Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications
        * Minor surgery within 1 months of the first dose of cabozantinib if therewere no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications.

In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery

* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the study agents. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients who require taking drugs that are strong inhibitors/inducers of CYP3A4 and cannot be switched to an alternative medication.

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-thecounter medicine or herbal product.

* Patients with greater than or equal to grade 2 peripheral neuropathy at baseline.
* The subject has had treatment with docetaxel for the treatment of metastatic castratesensitive prostate cancer within 6 months before the first dose of study treatment.
* The subject has had progression of prostate cancer during 6 cycles of prior docetaxel treatment for castrate sensitive disease.
* The subject has received chemotherapy for castration-resistant prostate cancer.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-09-07 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Dahut, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010 Sep-Oct;60(5):277-300. doi: 10.3322/caac.20073. Epub 2010 Jul 7. PMID 20610543
- [Background] Petrylak DP, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Berry D, Moinpour C, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1513-20. doi: 10.1056/NEJMoa041318. PMID 15470214
- [Result] A phase I and randomized phase II study of cabozantinib plus docetaxel and prednisone (C+DP) versus docetaxel and prednisone (DP) alone in metastatic castrate-resistant prostate cancer (mCRPC). Munjid Al Harthy, Ravi Amrit Madan, Fatima Karzai, Daniel Peter Petrylak, Joseph W. Kim, Philip M. Arlen, Marc Robert Theoret, Jenn Marte, Marijo Bilusic, Anna Couvillon, Guinevere Chun, Helen Owens, Amy Hankin, Lisa M. Cordes, William Douglas Figg, James L. Gulley, and William L. Dahut Journal of Clinical Oncology 2019 37:7_suppl, 173-173
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0204.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 participants were enrolled on this study. 4 participants were screen failures and were not assigned to any treatment groups. Data is shown for 45/49 participants. 13 participants were assigned to Ph II Arm A Docetaxel & Prednisone but only 12 started treatment; one participant declined to start treatment. Data is shown for 45/49 participants.
Groups:
- Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Cabozantinib: 20 mg by mouth (PO) everyday (QD); Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID)
- Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Cabozantinib: 40 mg by mouth (PO) everyday (QD); Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID)
- Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Cabozantinib: 60 mg by mouth (PO) everyday (QD); Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID)
- Ph II Arm A: Docetaxel + Prednisone: Cycle=21 days; Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg by mouth (PO) twice a day (BID)
- Ph II Arm B: Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID); Cabozantinib: 40 mg by mouth (PO) everyday (QD)
Period: Overall Study
Arm/Group | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone | Ph II Arm A: Docetaxel + Prednisone | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone
Started | 4 | 8 | 7 | 13 | 13
# of Patients Who Received Treatment | 4 | 8 | 7 | 12 | 13
Completed | 3 | 8 | 7 | 10 | 12
Not Completed | 1 | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Intercurrent illness | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone | Ph II Arm A: Docetaxel + Prednisone | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone | Total
Number analyzed (Participants) | 4 | 8 | 7 | 13 | 13 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 3 | 5 | 13
  >=65 years | 2 | 6 | 6 | 10 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.45 (11.67) | 66.16 (9.51) | 70.15 (12.03) | 67.72 (8.34) | 68.89 (8.46) | 67.34 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 4 | 8 | 7 | 13 | 13 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 4 | 8 | 6 | 12 | 10 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 3 | 5 | 6 | 18
  White | 3 | 5 | 3 | 8 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 8 | 7 | 13 | 13 | 45
Baseline Prostatic-Specific Antigen (PSA) [Median (Full Range); unit: ng/ml] — PSA normal range is 4 ng/ml or lower.
  ng/ml | 182.38 [0.01 to 508.5] | 73.71 [8.39 to 225] | 166.3 [2.06 to 897.9] | 346.9 [94.62 to 2649] | 65.6 [4.5 to 3940.38] | 118.4 [0.01 to 3940.38]
Prior Treatment with Enzalutamide or Abiraterone [Count of Participants; unit: Participants] | 3 | 5 | 4 | 8 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) of Cabozantinib + Docetaxel + Prednisone Compared to Docetaxel + Prednisone Alone
Description: PFS is the time interval from start of treatment to documented evidence of disease progression or death. Disease progression was assessed by the Response Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions as referenced by the smallest sum on study. Appearance of one or more new lesions on bone scan and/or two consecutive rising prostatic-specific antigen values above the baseline at a minimum of one week intervals. A normal PSA value is 4.0 ng/ml and lower.
Time Frame: From start date of treatment until the date of first documented progression, date of death from any cause and up to 40 months, whichever occurred first.
Population: Four participants came off study before restaging. One participant did not start treatment. Forty participants are evaluable for PFS. No participants received carbozantinib after progression from Docetaxel and Prednisone alone.
Measure: Median (Full Range); unit: months
Arm/Group | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone | Ph II Arm A: Docetaxel + Prednisone | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone
Number analyzed (Participants) | 3 | 8 | 7 | 10 | 12
months | 8 [2 to 39] | 13 [8 to 21] | 6 [2 to 13] | 10 [1 to 10] | 6.5 [2 to 24]

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the dose level at which no more than 1 of 6 patients experiences a dose limiting toxicity (DLT) at the level below that which had two instances of DLT. A DLT are defined as adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0) occurring during the first two cycles of therapy and related to the study medications (attributions: possible, probable, and definite) while fulfilling one of the following criteria: Any Grade 3 or greater non-hematologic toxicity except asymptomatic grade 3 hypertension, hypomagnesemia, hyponatremia, hypophosphatemia, hypocalcemia, and asymptomatic grade 4 uric acid. A treatment delay of > 2 weeks due to an adverse event (delays due to dental procedures are not included). Grade 4 neutropenia (absolute neutrophil count <500/µL lasting > 5 days. Febrile neutropenia. Grade 3 thrombocytopenia lasting for 7 days or more or thrombocytopenia < 50K/µL requiring platelet transfusion for bleeding.
Time Frame: First two cycles of treatment (each cycle is 21 days), approximately 42 days.
Population: Maximum tolerated dose was assessed only on phase 1 cohort participants. All 19 patients (e.g. 4 participants on dose level 1, 8 participants on dose level 2, and 7 participants on dose level 3) were included in the safety assessment to determine maximum tolerated dose.
Measure: Number; unit: mg
Groups:
- Ph I Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Cabozantinib: 20 mg, 40mg, and 60 mg by mouth (PO) everyday (QD); Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID)
Arm/Group | Ph I Cabozantinib + Docetaxel + Prednisone
Number analyzed (Participants) | 19
mg | 40

3. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events were assessed from the date treatment consent signed to date off study, approximately 45 months and 14 days for Arm A; 43 months and 14 days for Arm B; 9 months and 11 days for DL1; 27 months and 1 day for DL2; & 11 months & 25 days for DL3
Population: One participant in Arm A declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone | Ph II Arm A: Docetaxel + Prednisone | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone
Number analyzed (Participants) | 4 | 8 | 7 | 12 | 13
Participants | 4 | 8 | 7 | 12 | 13

4. Other Pre Specified Outcome: Number of Participants With a Dose Limiting Toxicities (DLTs)
Description: A DLT are defined as adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0) occurring during the first two cycles of therapy and related to the study medications (attributions: possible, probable, and definite) while fulfilling one of the following criteria: Any Grade 3 or greater non-hematologic toxicity except asymptomatic grade 3 hypertension, hypomagnesemia, hyponatremia, hypophosphatemia, hypocalcemia, and asymptomatic grade 4 uric acid. A treatment delay of > 2 weeks due to an adverse event (delays due to dental procedures are not included). Grade 4 neutropenia (absolute neutrophil count <500/µL lasting > 5 days. Febrile neutropenia. Grade 3 thrombocytopenia lasting for 7 days or more or thrombocytopenia < 50K/µL requiring platelet transfusion for bleeding.
Time Frame: First two cycles of treatment (each cycle is 21 days), approximately 42 days.
Population: DLT only pertains to DL1, 2 and 3. Arms A and B did not evaluate for DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Ph I Dose Level 1: Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Cabozantinib: 20mg by mouth (PO) everyday (QD); Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID)
- Ph I Dose Level 2: Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Cabozantinib: 40mg by mouth (PO) everyday (QD); Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID)
- Ph I Dose Level 3: Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Cabozantinib: 60mg by mouth (PO) everyday (QD); Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg PO twice a day (BID)
Arm/Group | Ph I Dose Level 1: Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 2: Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 3: Cabozantinib + Docetaxel + Prednisone
Number analyzed (Participants) | 4 | 8 | 7
Participants
  Neutropenic fever | 0 | 0 | 1
  Palmar plantar erythroderma | 0 | 0 | 1

5. Other Pre Specified Outcome: Number of Participants Achieving Prostatic-Specific Antigen (PSA) Decline of 30% or 50% From Baseline
Description: PSA normal range is 4 ng/ml or lower. Participants with PSA decline of 30% or 50% is the measures for prostate cancer based on conventional reporting metrics.
Time Frame: up to 38 months
Population: One participant randomized to Arm A declined to participate before treatment started.
Measure: Count of Participants; unit: Participants
Groups:
- Ph II Arm A Docetaxel + Prednisone: Cycle=21 days; Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg by mouth (PO) twice a day (BID)
- Ph II Arm B: Cabozantinib + Docetaxel + Prednisone: Cycle=21 days; Docetaxel: 75 mg/m^2 intravenous (IV) over 60 min on day 1; Prednisone: 5 mg by mouth (PO) twice a day (BID); Cabozantinib: 40mg by mouth (PO) everyday (QD)
Arm/Group | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone | Ph II Arm A Docetaxel + Prednisone | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone
Number analyzed (Participants) | 3 | 8 | 7 | 12 | 13
Participants
  Decline in PSA>30% from baseline | 0 | 5 | 5 | 5 | 10
  Decline in PSA>50% from baseline | 0 | 5 | 4 | 3 | 9

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date treatment consent signed to date off study, approximately 45 months and 14 days for Arm A; 43 months and 14 days for Arm B; 9 months and 11 days for Dose Level 1; 27 months and 1 day for Dose Level 2; and 11 months and 25 days for Dose Level 3.
Description: One participant in Arm/Group A declined to participate before treatment started.
Arm/Group | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone | Ph II Arm A: Docetaxel + Prednisone | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8 | 2/7 | 0/12 | 1/13
Serious Adverse Events (participants affected / at risk) | 2/4 | 5/8 | 2/7 | 3/12 | 3/13
Other Adverse Events (participants affected / at risk) | 4/4 | 8/8 | 7/7 | 12/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone (N=4) | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone (N=8) | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone (N=7) | Ph II Arm A: Docetaxel + Prednisone (N=12) | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ph I Dose Level 1:Cabozantinib + Docetaxel + Prednisone (N=4) | Ph I Dose Level 2:Cabozantinib + Docetaxel + Prednisone (N=8) | Ph I Dose Level 3:Cabozantinib + Docetaxel + Prednisone (N=7) | Ph II Arm A: Docetaxel + Prednisone (N=12) | Ph II Arm B: Cabozantinib + Docetaxel + Prednisone (N=13)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 2 (2) | 3 (3) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (11) | 1 (1) | 4 (5) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 3 (3) | 3 (3) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (3) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (3) | 6 (9) | 2 (3) | 3 (3) | 5 (7)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 3 (4) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 5 (5) | 2 (3) | 6 (8) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (12) | 5 (6) | 1 (9) | 1 (1) | 1 (2)
Infusion related reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 1 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 4 (4)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (8) | 4 (5) | 2 (2) | 4 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Extraosseous extension
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 4 (4) | 2 (6) | 4 (4) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 1 (5)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Vascular disorders - Other, peripheral vascular disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 4 (6) | 2 (3) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Weight loss (Investigations) | 0 (0) | 6 (10) | 2 (2) | 1 (1) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7) | 3 (3) | 0 (0) | 8 (8)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 6 (11) | 3 (5) | 0 (0) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (3) | 0 (0) | 4 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (26) | 3 (4) | 0 (0) | 6 (8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, skin discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 4 (14)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Burning sensation in legs/bones
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (7) | 7 (16) | 4 (6) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, dermatitis-eye (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 5 (8) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (4) | 3 (8) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, vasculopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, R. thigh lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, dermatitis-hand (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT01683994/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT01683994/ICF_001.pdf